CLINICAL TRIAL: NCT04465318
Title: Electronic Cigarettes as a Harm Reduction Strategy Among Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-00839
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: COPD
Keywords: E-cigarettes
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Vaping | interventions — Electronic Nicotine Delivery Systems; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-cigarettes (EC) (Experimental): EC + Counseling
  Interventions: Other: E-cigarette (EC); Behavioral: Smoking Harm Reduction Counseling Sessions
- Nicotine Replacement Therapy (NRT) (Active Comparator): NRT + Counseling
  Interventions: Other: Nicotine Replacement Therapy (NRT); Behavioral: Smoking Harm Reduction Counseling Sessions

INTERVENTIONS:
Other: E-cigarette (EC) — NJOY Daily E-cigarettes are self-contained and non-refillable. Each DAILY provides approximately 300 puffs, comparable to a full pack of cigarettes.
  Arms: E-cigarettes (EC)
Other: Nicotine Replacement Therapy (NRT) — Participants in the NRT arm will receive 21 mg nicotine patch (for those with CPD >= 20) or 14 mg nicotine patch (for those with CPD < 20) + 4 mg nicotine gum. CPD stands for Cigarettes Per Day.
  Arms: Nicotine Replacement Therapy (NRT)
Behavioral: Smoking Harm Reduction Counseling Sessions — Counseling will cover health education, social support issues, and motivational enhancement to improve self-efficacy while addressing other aspects know to contribute to smoking among people with COPD (e.g., tips on dealing with depression)

SUMMARY:
The study team proposes a two-arm pilot study randomizing participants with COPD who smoke combustible cigarettes (CC) to counseling + NRT (standard of care) or counseling + e-cigarettes.

DETAILED DESCRIPTION:
Globally, chronic obstructive pulmonary disease (COPD) is projected to be the third largest cause of death by 2030 and in the US over 16 million people have COPD. Smokers are four and a half times more likely to develop COPD than non-smokers, with the likelihood of COPD increasing progressively with the duration and intensity of smoking. Among those with COPD, smoking cessation is the most effective means of slowing the decline of lung function and overall disease progression. Patients at all stages of COPD benefit from quitting smoking. Over 90% of COPD deaths occur in current smokers, however 47.1% of people with COPD continue to smoke. Electronic cigarettes (E-cigarettes) could help people reduce the harm of combustible cigarettes (CC) through reductions in number of Cigarettes per Day (CPD) or quitting CC completely by addressing both nicotine and behavioral dependence. Although there are associated health risks, all available evidence indicates that E-cigarettes are safer than CC. Unlike CC, e-cigarettes are not associated with coronary heart disease or myocardial infarction. The purpose of this mixed methods study is to identify barriers and facilitators, as well as to assess preliminary effectiveness of e-cigarettes as a harm reduction strategy among people with COPD.

ELIGIBILITY:
Inclusion Criteria:

1. an ambulatory ICD-10 code for COPD in the last 12 months and a COPD Assessment Tool (CAT) score on the screening ≥10.
2. ages 21-75 (the legal age for purchasing e-cigarettes is 21)
3. current CC smokers (more than 5 packs in a lifetime; smokes 4 or more days/week)
4. smokes at least 10 cigarettes per day on days they smoke CC
5. motivated to quit smoking (at least a 5 on a 10-point Likert scale)
6. Participants must be able to provide consent, agree to be randomized and followed-up with, a working telephone number and/or a system with teleconferencing capabilities (e.g. smartphone or computer), a phone with text messaging capabilities, and be willing to use an e-cigarette or NRT for 12 weeks. To reduce attrition, participants will be asked to provide one additional contact as a backup for follow up on appointments.

Exclusion Criteria:

1. A CAT score >30 representing severe COPD
2. are pregnant (as determined by urine pregnancy test for women under age 52) or breastfeeding (self-reported). Women of childbearing age must also be willing to use an approved form of birth control during the course of the study if not practicing abstinence. Approved birth control methods include: hormonal birth control (e.g. "the pill"), barrier methods (e.g. condoms, diaphragm), and intrauterine devices (IUDs).
3. diagnosis of any medical condition (unstable angina/heart disease) or psychiatric condition precluding use of nicotine patch or gum as determined by the MD of this study, Dr. Scott Sherman (NYS license #171632), or by the subject's primary care doctor.
4. reporting using NRTs or e-cigarettes within the last 30 days

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Number of participants who achieve 50% reduction in Cigarettes Per Day (CPD) | 12 weeks
  Smoking reduction will be measured by a self-report.
Average change in score on the mMRC Dyspnea Scale | Baseline, 12 weeks
  The mMRC Dyspnea Scale is a self-rating tool that quantifies disability attributable to breathlessness. The score ranges from 0 to 4. The higher the score, the higher the disability of breathlessness poses on day-to-day activities.

SECONDARY OUTCOMES:
Number of participants who reported satisfaction with use of e-cigarettes | 12 weeks
Number of participants who reported additional use of tobacco products and/or marijuana | 12 weeks
Change in score of COPD Assessment Test (CAT) | Baseline, 12 weeks
  CAT consists of 8 statements, each scored between 0-5 for a total score range of 0-40. The higher the score, the worse the COPD symptoms.
Change in score of Clinical COPD Questionnaire (CCQ) | Baseline, 12 weeks
  CCQ consists of 10 questions, each scored between 0-6 for a total score range of 0-60. The higher the score, the worse the COPD symptoms and more limitations due to the COPD symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Scott E. Sherman, MD, MPH, Principal Investigator — NYU Langone Health; Elizabeth Stevens, PhD, MPH, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to scott.sherman@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Rojas SV, Kyanko KA, Wisniewski R, O'Connor K, Li R, Xiang G, Vojjala M, Wilker O, Sherman SE, Stevens ER. Patient perceptions of the use of e-cigarettes in smoking treatment programs: a qualitative analysis. Addict Sci Clin Pract. 2025 May 30;20(1):45. doi: 10.1186/s13722-025-00575-w. PMID 40442834
- [Derived] Stevens ER, Lei L, Cleland CM, Vojjala M, El-Shahawy O, Berger KI, Kirchner TR, Sherman SE. Electronic cigarettes as a harm reduction strategy among patients with COPD: protocol for an open-label two arm randomized controlled pilot trial. Addict Sci Clin Pract. 2022 Jan 6;17(1):2. doi: 10.1186/s13722-021-00284-0. PMID 34991693